CLINICAL TRIAL: NCT01255813
Title: Sphenopalatine Ganglion Stimulation for the Acute Treatment of Cluster Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Autonomic Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pathway CH-1 (CIP-001)
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Cluster Headache
Keywords: Chronic Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Other: Control
- Sub-perception (Experimental)
  Interventions: Device: Stimulation (Sub-perception)
- Full Stimulation (Experimental)
  Interventions: Device: Stimulation (Full)

INTERVENTIONS:
Device: Stimulation (Sub-perception) — Stimulation applied below the perception threshold
  Arms: Sub-perception
Device: Stimulation (Full) — Stimulation applied above the perception threshold
  Arms: Full Stimulation
Other: Control — No stimulation applied
  Arms: Placebo

SUMMARY:
The purpose of the proposed clinical study is to evaluate the use of an implanted Neurostimulator to provide Sphenopalatine Ganglion (SPG) stimulation for the management of the pain associated with cluster headaches.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years old (inclusive).
* Subject has been diagnosed with chronic cluster headache according to the 2004 International Headache Society (IHS) criteria 3.1.2.
* Subject reports a minimum of 4 cluster headaches per week.
* Subject reports dissatisfaction with current cluster headache treatment (Criterion includes both preventive or abortive therapy per the Investigator's standard of care. Reasons for dissatisfaction with existing headache therapies may include failure of therapies, contraindication, side effects of therapies, or patient refusal of available therapies)
* Subject is able to distinguish cluster headaches from other headaches (i.e., tension-type headaches).
* Subject has the ability to read and comprehend, and to reliably record information as required by the Protocol.
* Subject is able to provide written informed consent prior to participation in the study.

Exclusion Criteria:

* Subject has had a change in type or dosage of prophylactic headache medications < one (1) month prior to study enrollment
* Subject has undergone facial surgery in the area of the pterygopalatine fossa or zygomaticomaxillary buttress ipsilateral to the planned implant site within the last four (4) months.
* Subject has active oral or dental abscess.
* Subject has been treated with radiation to the facial region within the last six (6) months.
* Subject has been diagnosed with any major infectious processes such as osteomyelitis, or primary or secondary malignancies involving the face that have been active or required treatment in the past six (6) months.
* Subject has other significant pain problem that might confound the study assessments in the opinion of the Investigator.
* Subject is a woman of childbearing age who is pregnant, nursing, or not using contraception.
* Subject is currently participating or has participated in the last month in another clinical study in which the subject has, is, or will be exposed to an investigational or non-investigational drug or device.
* Subject is felt to be at risk of non-compliance (e.g., for completing the diary or maintaining a stable headache medicine regimen) in the Investigator's opinion.
* Subject has had previous lesional radio-frequency ablation of the ipsilateral sphenopalatine ganglion (SPG).
* Subject has had blocks of the ipsilateral SPG in the last three (3) months.
* Subject has undergone botulinum toxin injections of the head and/or neck in the last three (3) months.
* Subject has or requires a pacemaker/defibrillator or other implantable device having a sense amplifier.
* Subject has a history of bleeding disorders or coagulopathy or is unable to discontinue anticoagulation, antiplatelet, or GP IIb IIIa inhibitor medication in preparation for the implantation procedure.
* Subject is not suitable for the study for any reason in the judgment of the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of device related Serious Adverse Events (SAEs) | Implant through the Experimental Period
Acute Pain Relief response (as defined by patient) | 15 minutes

SECONDARY OUTCOMES:
Pain Freedom | 15 minutes
Rescue medication use | 90 minutes
  Use of medications to treat headache pain within 90 minutes after initiating therapy.
Pain Relief after initiating therapy | 30 minutes
Pain Relief after initiating therapy | 60 minutes
Pain Relief after initiating therapy | 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jean Schoenen, M.D., Principal Investigator — Professor of Functional Neuroanatomy, Leige University
Locations (5):
- Citadelle Hospital, Liège, Belgium
- Danish Headache Center, Dept. of Neurology, Glostrup Hospital, Glostrup Municipality, Denmark
- Germany (2):
  - Headache Center, Dept. of Neurology, University Duisburg-Essen, Essen
  - Institut fur systemische Neurowissenschaften, Universitastsklinikum Hamburg-Eppendorf (UKE), Hamburg
- Department of Neurology, University Clinic Hospital, University of Valencia, Valencia, Spain